CLINICAL TRIAL: NCT06696040
Title: Immediate Effects of Mobilization Performed by Passive Kinesiotherapy Equipment on Lower Limbs on Spasticity and Gait in Neurological Patients
Brief Title: Immediate Effects on Gait and Spasticity After the Use of Passive Kinesiotherapy Equipment in the Lower Limbs of Neurological Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fernanda Trubian (Other)
Responsible Party: Sponsor-Investigator, Fernanda Trubian, PhD student in Health Sciences, Universidade de Caxias do Sul
Organization: Universidade de Caxias do Sul (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 83118724.0.0000.5341
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-11

CONDITIONS: Hemiparesis; Paraparesis; Tetraparesis; Cerebral Palsy; Spastic Gait; Spasticity
Keywords: Gait; Spasticity; Passive Kinesiotherapy; Spastic Gait; Passive mobilization device
MeSH Terms: conditions — Paresis; Paraparesis; Quadriplegia; Cerebral Palsy; Gait Disorders, Neurologic; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre-intervention and immediate post-intervention (Experimental)
  Interventions: Device: Passive mobilization using a device

INTERVENTIONS:
Device: Passive mobilization using a device — The protocol consists of three moments: initial assessment, use of the device, and final assessment.
  In the initial assessment, participants will be positioned supine on a stretcher, where the muscle tone of the lower limb(s) will be tested using the Modified Ashworth Scale. After the physical test with the Modified Ashworth Scale, the TUG test will be carried out, and, finally, gait assessment with the BAIOBIT Inertial Meter with Accelerometer and Gyroscope.
  At the end of the initial assessment, the Autofisio500 device will be used. To do this, the participant will be positioned again and comfortably supine on the stretcher, and the previously tested lower limb will be attached to the device for movement, between the knee and ankle joints, for 30 minutes, at maximum speed (11 RPM).
  For the final assessment, the Modified Ashowrth Scale, TUG and gait assessment with the Inertial Meter with Accelerometer and BAIOBIT Gyroscope will be applied again.

SUMMARY:
Undergo assessment of muscle tone (Ashworth Scale), gait (BAIOBIT) and risk of falling (Timed Up and Go) before using the device; Use the device on the spastic lower limb(s) for 30 minutes; Go through the same assessment carried out previously.

ELIGIBILITY:
Inclusion Criteria:

* agree and sign the Free and Informed Consent Form or signature of the person responsible
* individuals with spasiticity (hemiparetic, paraparetic, tetraparetic and hemiparetic children with cerebral palsy)

Exclusion Criteria:

* over 18 years old whose ability to sign the Free and Informed Consent Form is compromised, or who understand it, but are not responsible for signing the Free and Informed Consent Form
* present cardiovascular, neurological, musculoskeletal instability or other condition(s) that interfere with the use or positioning of the device or gait assessment
* present cognitive deficits that interfere with understanding the ICF and/or understanding how to carry out the protocol
* For the children's group, participants who: 1) are under 8 years of age and/or over 13 years of age will be excluded; 2) no person responsible for signing the TCLE; 3) present cognitive deficits that interfere with understanding the ICF and/or understanding how to carry out the protocol

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Gait kinematics | Immediate post-evaluation (after using the device for 30 minutes)
  Assessment of gait kinematics using the BAIOBIT pre and post intervention

SECONDARY OUTCOMES:
Muscle tone - spasticity | Immediately after using the device for 30 minutes
Timed Up and Go | Immediately after using the device for 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade de Caxias do Sul, Caxias Do Suk, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Participants in this study will have their identities preserved, information from this research will be treated confidentially and confidentially by the responsible researchers and their direct collaborators. All data will be made anonymous (that is, it will only contain your participation number in the study, but not your name) and only these researchers will be able to handle this database. This ensures the privacy and confidentiality of participant data in any publication of results.
  The data will be stored in a file, under the custody of the responsible researcher, for 5 (five) years, containing individual files.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- See also: Feasibility and safety of early lower limb robot-assisted training in sub-acute stroke patients: a pilot study — https://pubmed.ncbi.nlm.nih.gov/28084064/
- See also: Feasibility and outcomes of supplemental gait training by robotic and conventional means in acute stroke rehabilitation — https://pubmed.ncbi.nlm.nih.gov/37794474/
- See also: Effects of aerobic cycling training on mobility and functionality of acute stroke subjects: A randomized clinical trial — https://pubmed.ncbi.nlm.nih.gov/33386826/
- See also: Enhanced Gait-Related Improvements After Therapist- Versus Robotic-Assisted Locomotor Training in Subjects With Chronic Stroke A Randomized Controlled Study — https://pubmed.ncbi.nlm.nih.gov/18467648/